CLINICAL TRIAL: NCT02737254
Title: The Effect of Oxytocin on the Training of Attachment-related Interpretation Bias in Middle Childhood
Brief Title: Oxytocin and Attachment-related Interpretation Bias
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: S57012; 2014-005352-25 (EudraCT Number)
Record Dates: First submitted 2016-03-23; First posted 2016-04-13 (Estimated); Last update posted 2016-11-08 (Estimated); Status verified 2016-02

CONDITIONS: Trust
Keywords: Attachment; Oxytocin; Cognitive bias modification; Middle childhood
MeSH Terms: interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Oxytocin and Secure CBM training (Experimental)
  Interventions: Drug: Oxytocin; Other: Secure CBM training
- Placebo and Secure CBM training (Active Comparator)
  Interventions: Drug: Placebo; Other: Secure CBM training
- Oxytocin and Neutral CBM training (Active Comparator)
  Interventions: Drug: Oxytocin; Other: Neutral CBM training
- Placebo and Neutral CBM training (Placebo Comparator)
  Interventions: Drug: Placebo; Other: Neutral CBM training

INTERVENTIONS:
Drug: Oxytocin — 40 IU/ML nasal spray. One administration: children <40kg administer 12IU, children >40kg administer 24IU.
  Arms: Oxytocin and Neutral CBM training; Oxytocin and Secure CBM training
Drug: Placebo — NaCl 0,9 % nasal spray.
  Arms: Placebo and Neutral CBM training; Placebo and Secure CBM training
Other: Secure CBM training — Children are trained to interpret ambiguous maternal behavior in a secure way.
  Arms: Oxytocin and Secure CBM training; Placebo and Secure CBM training
Other: Neutral CBM training — Children receive a training unrelated to the interpretation of maternal behavior.
  Arms: Oxytocin and Neutral CBM training; Placebo and Neutral CBM training

SUMMARY:
The purpose of this study is to investigate the effects of oxytocin and a cognitive bias modification (CBM) procedure on children's trust in their mother.

DETAILED DESCRIPTION:
Previous research has shown that children can be trained to interpret ambiguous interactions with mother in a more secure way by use of a CBM procedure. A secure attachment-related processing bias can causally increase children's trust in mother's availability. The present study tests whether intranasal administration of oxytocin can increase the effect of a secure cognitive bias training. Oxytocin is a neuropeptide that is involved in human attachment and bonding. Intranasal administration of oxytocin can increase trust among people. After oxytocin or placebo administration, children are either trained to interpret ambiguous interactions with mother in a secure way or receive a neutral training unrelated to interpretation of maternal behavior. Pre- and post-intervention children's trust in mother, support seeking behavior and interpretation of maternal behavior is assessed. Moreover, possible oxytocin side-effects will be monitored.

ELIGIBILITY:
Inclusion Criteria:

* Between 8 and 13 years old
* Mother can also participate

Exclusion Criteria:

* Known oxytocin allergy
* Currently using medication
* Kidney or cardial condition

Ages: 8 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2016-03; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Change in trust in mother | Immediately before and immediately after intervention
  Trust in mother as measured by People in My Life Trust subscale.

SECONDARY OUTCOMES:
Change in attachment-related behavior towards mother | Immediately before and immediately after intervention
  Observation of the quality of the approach of child towards mother during a puzzle task.
Change in secure interpretation of ambiguous maternal behavior | Immediately before and immediately after intervention
  After reading scenarios describing ambiguous maternal behavior, children will be presented with sentences describing secure interpretations of this behavior and are asked to rate on a 4-point Likert scale to what extent this did or did not happen in the scenario. Thereby, children's spontaneous secure interpretation of ambiguous maternal behavior can be assessed.
Change in insecure interpretation of ambiguous maternal behavior | Immediately before and immediately after intervention
  After reading scenarios describing ambiguous maternal behavior, children will be presented with sentences describing insecure interpretations of this behavior and are asked to rate on a 4-point Likert scale to what extent this did or did not happen in the scenario, assessing children's spontaneous insecure interpretation of ambiguous maternal behavior.
Interpretation speed of positive maternal behavior | Throughout the CBM training, from around 60 minutes until 110 minutes after the start of the procedure
  Reaction times to scenarios describing secure maternal behavior.
Interpretation speed of negative maternal behavior | Throughout the CBM training, from around 60 minutes until 110 minutes after the start of the procedure
  Reaction times to scenarios describing insecure maternal behavior.

OTHER OUTCOMES:
Oxytocin side-effects | Immediately after intervention and 24 hours after intervention
  Questionnaire on possible oxytocin side-effects.
Change in mood | Immediately before nasal spray, immediately before CBM training and immediately after CBM training
  Children rate on two visual analogous scales how happy and how sad they feel.

CONTACTS AND LOCATIONS:
Overall Officials: G. Bosmans, Prof. dr., Principal Investigator — KU Leuven
Locations (1):
- KU Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Verhees MWFT, Ceulemans E, Bakermans-Kranenburg MJ, van IJzendoorn MH, de Winter S, Bosmans G. The effects of Cognitive Bias Modification training and oxytocin administration on trust in maternal support: study protocol for a randomized controlled trial. Trials. 2017 Jul 14;18(1):326. doi: 10.1186/s13063-017-2077-2. PMID 28709470